CLINICAL TRIAL: NCT05495646
Title: Infection Related to Short-term Central Venous Catheters: an Observational Study in Surgical Patients
Brief Title: Infection Related to Short-term Central Venous Catheters
Status: Completed | Type: Observational
Sponsor: Ángel Becerra (Other)
Responsible Party: Sponsor-Investigator, Ángel Becerra, Principal Investigator, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Other Study IDs: 150030
Record Dates: First submitted 2022-08-05; First posted 2022-08-10 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Catheter-Related Infections
MeSH Terms: conditions — Catheter-Related Infections | interventions — Catheterization, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Central catheter insertion — The data will be obtained through the review of the medical records and the clinical follow-up of each patient to evaluate the technique of inserting the device, the possible risk factors of catheter-related infection, its clinical manifestations and the data microbiological.

SUMMARY:
This study aims to evaluate the incidence of infection of short-term central venous catheters by comparing different cannulation techniques (by anatomical references and under ultrasound control) and according to the experience of the operator in patients undergoing elective surgery.

A prospective observational study will be carried out in which all scheduled surgery patients who have a central venous line inserted for 12 months will be included. Those under 18 years of age, patients with catheters lasting more than 14 days and those who do not sign the informed consent will be excluded from this study. A chest X-ray will be performed on all patients in order to diagnose possible complications associated with the technique and, only in case of suspected infection, culture of the catheter tip and blood cultures of blood obtained from the catheter and peripheral blood will be requested.

DETAILED DESCRIPTION:
A prospective observational study will be carried out. The maximum time between the intervention and the final evaluation will be 21 days, since the study evaluates the infection related to short-term catheters and its probable improvement after the removal of the device.

All patients undergoing elective surgery who have a central venous line inserted for 12 months will be included in the study. Those under 18 years of age, patients with catheters lasting more than 14 days and those who do not sign the informed consent will be excluded.

A follow-up of the central venous catheters that are inserted in those patients scheduled for surgery who have an indication for it will be carried out. The criteria for choosing the access route will be carried out according to the usual clinical practice of the responsible anesthesiologist.

The asepsis measures that will be carried out both in the insertion and in the maintenance of the catheter will be those used on a regular basis, which follow the recommendations of the guidelines for the prevention of infections related to intravascular catheters of the American Center for Control and Prevention. of Diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgery who have a central venous line inserted during the three months in which the study runs

Exclusion Criteria:

* Patients under 18 years of age
* Patients who need to wear the central venous catheter for more than 14 days
* Patients who do not sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery during the three months in which the study is carried out who need a central venous catheter.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Incidence of infection among short-term central venous catheters inserted in the scheduled perioperative setting. | From the immediate postoperative period to the 21st postoperative day
  Review of the clinical follow-up of each patient to evaluate the appearance of catheter related infection through its clinical manifestations and microbiological data.

SECONDARY OUTCOMES:
Number of patients suffering from complications after the different techniques and operators. | From the immediate postoperative period to the first postoperative day
  Review of the clinical follow-up of each patient to evaluate the technique of inserting the central venous catheter.
Assess risk factors for catheter-related infection | From the immediate postoperative period to the 21st postoperative day
  Review of the medical records and the clinical follow-up of each patient to evaluate the risk factors for suffering from catheter-related infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Ángel Becerra, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Undecided